CLINICAL TRIAL: NCT06490185
Title: Clinical Significance of Peri-appendiceal Abscess and Phlegmon in Acute Complicated Appendicitis Patients Undergoing Emergency Appendectomy: A Single-center Retrospective Study
Brief Title: Peri-appendiceal Abscess and Phlegmon in Acute Complicated Appendicitis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhongshan-HHY-06
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Acute Complicated Appendicitis With Peri-appendiceal Abscess or Phlegmon
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical data collection — Clinical significance of peri-appendiceal abscess and phlegmon in acute complicated appendicitis patients undergoing emergency appendectomy

SUMMARY:
This study aim to analyze the clinical data of patients who underwent emergency appendectomy for acute complicated appendicitis with peri-appendiceal abscess or phlegmon, identify factors influencing the post-operative length of hospital stay (LOS), and improve treatment strategies.

DETAILED DESCRIPTION:
Appendicitis is defined as inflammation of the vermiform appendix and worldwide is the most common reason for emergency abdominal surgery. Globally, the annual incidence is 96.5 to 100 cases per 100 000 adult population. For acute uncomplicated appendicitis, antibiotic therapy has emerged as the primary treatment, often allowing patients to avoid surgery. However, the management of acute complicated appendicitis requires careful consideration of various treatment options.

Complicated appendicitis, characterized by peri-appendiceal phlegmon or abscess formation, presents additional challenges and often requires a more comprehensive treatment approach. Management strategies have evolved to incorporate both conservative and surgical treatments, tailored to the patient's condition. Typically, for early-stage appendicitis (duration of symptoms ≤72 hours) with peri-appendiceal phlegmon, surgical treatment is recommended, while late-stage appendicitis (duration of symptoms >72 hours) or cases with peri-appendiceal abscess formation are initially managed conservatively with percutaneous drainage and antibiotics. Despite this, some patients still prefer surgical intervention for various reasons. Currently, there is a lack of studies on the outcomes of patients with acute complicated appendicitis who opt for surgery over conservative treatment, highlighting the need for further research.

In practical terms, the benefits and risks of all treatment options should be thoroughly presented and discussed. Recommendations for surgery versus a conservative treatment-first approach should be based on individual clinical and radiographic findings, as well as patient treatment expectations and preferences. This study aim to investigate the clinical significance of peri-appendiceal abscess or phlegmon in the surgical management of acute complicated appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were aged ≥18 years, Patients who were clinically diagnosed with acute appendicitis, Patients who had a peri-appendiceal abscess or phlegmon on CT scan, Patients who opted to undergo immediate emergency surgery as their primary choice, Patients who refused conservative treatment first (antibiotic therapy and ultrasound/CT-guided drainage).

Exclusion Criteria:

* Patients younger than 18 years, Patients have a history of prior malignancies, Patients with diffuse peritonitis, Patients with incomplete clinical or pathological records.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute complicated appendicitis patients with peri-appendiceal abscess or phlegmon who met the criteria.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The post-operative length of hospital stay (LOS) | January 01, 2025 to December 31, 2025.